CLINICAL TRIAL: NCT05971901
Title: A Combinatorial Biomarker for Infection Diagnosis in Children
Acronym: CROCODILE-I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Cihan Papan, Principial Investigator, Universität des Saarlandes
Other Study IDs: 233/22
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Tract Infections; Fever
MeSH Terms: conditions — Respiratory Tract Infections; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BV use cases: cases in whom BV was ordered
  Interventions: Diagnostic Test: BV
- BV non-use cases: cases in whom BV was not ordered

INTERVENTIONS:
Diagnostic Test: BV — The use of the BV test, ordered at the discretion of the treating physician
  Groups: BV use cases

SUMMARY:
To describe the epidemiology, clinical presentation, diagnosis, therapy, and treatment outcomes of patients in whom the combination biomarker BV (combination of TRAIL, IP-10, and CRP) is used, and to compare them with control patients without BV measurement.

Secondary objectives:

* Qualitative evaluation of indication as well as adherence to the test result.
* Comparison of antimicrobial therapy, performed diagnostics, hospitalization, and outcomes between patients with high BV score (bacterial) and patients with low BV score (viral).

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of acute bacterial or viral infection
* Requirement of at least one BV test during medical presentation

Exclusion Criteria:

* lack of informed consent

Min Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients for whom the treating physicians request the determination of the BV score from the patient's serum due to a suspected infection can be included in this study, provided that they meet the above inclusion criteria, are capable of giving consent and agree to participate in the study (or, in the case of incapacitated patients, written consent is obtained from their legal guardian, health care proxy or custodian).
Sampling Method: Non-Probability Sample
Enrollment: 770 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Antibiotics | up to 30 days
  Number of participants treated with antibiotics

SECONDARY OUTCOMES:
Antibiotic duration | up to 30 days
  Length of antibiotic treatment per participant
Hospitalization | up to 30 days
  Number of participants admitted to the hospital
Complications | up to 30 days
  Rate of complications per participant
Tests | up to 30 days
  Rate of ancillary tests per participant

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Papan, MD, Principal Investigator — Universität des Saarlandes
Locations (4):
- Germany (4):
  - Sana Kliniken, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Saarland University, Homburg
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided